CLINICAL TRIAL: NCT00476814
Title: Cystic Fibrosis Transmembrane Conductance Regulator Function as Measured by Nasal Potential Difference Measurements in Patients With Primary Sclerosing Cholangitis
Brief Title: NPD Measurements in PSC Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: will002-HMO-CTIL
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: cystic fibrosis,; nasal potential difference,; primary sclerosing cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing; Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Sclerosing Cholangitis (PSC) is a chronic disorder of the liver causing jaundice and liver damage. When Cystic Fibrosis affects the liver, the damaged liver looks like the liver in PSC. This study is designed to answer the question whether isolated PSC may be a form of CF only in the liver

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is a progressive autosomal recessive disorder caused by defects in the cystic fibrosis transmembrane conductance regulator gene (CFTR). CFTR mutations cause loss or impairment of CFTR-mediated ion transport across epithelial cell membranes. CF affects many organs including the respiratory tract, pancreas, intestine, liver and the male reproductive tract. Liver disease occurs less frequently than pulmonary disease. CFTR is expressed in the bile duct epithelial cells and is responsible for the hydration of biliary secretions.

CF was until recently, thought to be a multi-organ disease. However, there are now recognized non-classical presentations of CF involving a few organs only and now there is well established data on single -organ involvement including Congenital Absence of the Vas Deferens and recurrent pancreatitis.

CF and PSC have several features in common. They both affect intrahepatic bile ducts by inspisated biliary secretions, chronic inflammation and fibrosis. Is PSC the "single-organ presentation" of CF? Patients with PSC will undergo testing of the CF protein channel by nasal potential testing. This test is performed by insering a thin plastic tube 2 to 3 cms into the nostril and chloride transport can be measured. This test may shows that the patient has an abnormality in the CF protein channel.

ELIGIBILITY:
Inclusion Criteria:

* Age > 10 years
* Patients diagnosed as Non-IBD PSC
* Patients diagnosed as IBD PSC

Exclusion Criteria:

* Age < 10 years

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wilschanski, Dr, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel